CLINICAL TRIAL: NCT00551837
Title: Immune Response to Influenza Vaccination
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-12-14
Record Dates: First submitted 2007-10-30; First posted 2007-10-31 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Solid Organ Transplantation; Chronic Kidney Disease
Keywords: Lung Transplantation; Kidney Transplnatation; Chroinic Kidney Disease; Influenza
MeSH Terms: conditions — Renal Insufficiency, Chronic; Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to evaluate the immune response to a routine influenza vaccination. Influenza vaccination is given as part of routine standard of care in these individuals and is not part of the study protocol. The study will evaluate for a change in response to common antigens over time after influenza vaccination to determine if changes are related to the development of chronic rejection after solid-organ transplantation. We hypothesize that the influenza vaccine contributes to the alloreactivity of T cells verses common HLA types in the donor pool.

ELIGIBILITY:
Inclusion Criteria:

* Transplant recipients (lung or kidney) 18 years or older, more than 3 months after transplantation
* Transplant candidates (kidney) 18 years or older, to recieve influenza vaccination
* Healthy volunteers to receive influenza vaccination

Exclusion Criteria:

* Under 18 years of age
* Pregnant
* Medical contraindication for vaccine
* Transplant recipients receiving acute rejection therapy within one month
* Healthy volunteers with autoimmune disease or medications to mediate immune function
* Receipt of live, attenuated influenza vaccine, instead of injectable vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Lung and kidney transplant recipients, patients with chronic kidney disease and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2006-11; Primary Completion 2008-04 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Poggio, MD, Study Director — The Cleveland Clinic